CLINICAL TRIAL: NCT07381465
Title: Efficacy and Safety of IL-1 Inhibitors in the Treatment of Mild to Moderate Systemic Lupus Erythematosus With Inadequate Response to Conventional Therapy: A Single-Centre, Single-Arm, Pilot Study
Brief Title: Efficacy and Safety of IL-1 Inhibitors in Mild to Moderate Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTAR012
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Firsekibart group (Experimental): Firsekibart combined with standard therapy: subcutaneous injection of 200mg Firsekibart at weeks 0, 4 and 8. Firsekibart monotherapy discontinued at weeks 12-24, with all other standard treatments unchanged. Observe for recurrence; if recurrence occurs, patients will be removed from the group and receive additional therapy.
  Interventions: Drug: Firsekibart

INTERVENTIONS:
Drug: Firsekibart — Firsekibart combined with standard therapy: subcutaneous injection of 200mg Firsekibart at weeks 0, 4 and 8. Discontinue Firsekibart at weeks 12-24, with all other standard treatments unchanged. Observe for recurrence; if recurrence occurs, patients will be removed from the group and receive additional medication.

SUMMARY:
Systemic lupus erythematosus (SLE) is a systemic autoimmune disorder in which pro-inflammatory factors of the IL-1 family play a pivotal role in its pathogenesis. In SLE patients, an innate immune hyperreactivity coupled with excessive inflammasome activation leads to substantial IL-1β production, triggering inflammatory phenotypes such as fever and serositis. For SLE patients unresponsive to conventional therapies, particularly those exhibiting high fever and serositis indicative of innate immune overactivation, effective targeted treatments remain scarce. Firsekibart, as a first anti-IL-1β biologic, holds promise in delivering novel therapeutic benefits for SLE patients with high-inflammatory phenotypes who prove refractory to standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years, male or female; female participants must not be pregnant or breastfeeding and must agree to use effective contraception during the trial period.
* Meets the 2012 SLICC classification criteria for SLE or the 2019 ACR/EULAR classification criteria for SLE;
* Mild to moderate disease activity, 1 point ≤ SLEDAI ≤ 12 points (cSLEDAI ≠ 0);
* The presence of at least one of the following recent clinical manifestations: fever (excluding fever caused by infection, tumor, endocrine or metabolic disorders, central nervous system diseases, medications, or physical factors), serositis (such as pericarditis or pleurisy), arthritis, rash, or alopecia;
* ESR or CRP exceeds the upper limit of normal, i.e. ESR > 20 mm/h or CRP > 10 mg/L;
* Patients had received standard therapy prior to study drug administration: ≤1 immunosuppressive agent for at least 12 weeks (methotrexate ≤15 mg/week, azathioprine ≤100 mg/day, mycophenolate mofetil ≤1.5 g/day, tacrolimus ≤2 mg/day, cyclosporine ≤150 mg/day, sirolimus ≤1.5 mg/day); Hydroxychloroquine (HCQ) may be used; Patients previously treated with biologics (e.g., Belimumab, Telitacicept, Anifrolumab) with inadequate response may also be considered for inclusion, provided they undergo a washout period of three half-lives during screening.
* The patient voluntarily participated in this trial, demonstrated good compliance, and possessed the capacity to understand and sign the informed consent form prior to the study.

Exclusion Criteria:

* SLE with major organ dysfunction, including impaired consciousness, cognitive decline, renal insufficiency, cardiac insufficiency (NYHA class 3 or 4), pulmonary hypertension, and pulmonary interstitial disease.
* Active SLE organ involvement, including but not limited to active lupus encephalopathy, active lupus nephritis (proteinuria ≥1g/24h), cardiac involvement, gastrointestinal involvement, diffuse alveolar haemorrhage, thrombocytopenic purpura, hemophagocytic syndrome, and retinopathy.
* SLE coexisting with other autoimmune diseases potentially affecting efficacy assessment, including but not limited to rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, and psoriasis.
* Abnormal liver function: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times the upper limit of normal; total bilirubin (TBIL) > 1 times the upper limit of normal.
* Any active malignancy or history of malignancy within the preceding five years.
* Concurrent conditions requiring glucocorticoid therapy, such as asthma or Crohn's disease.
* Acute or chronic infections requiring anti-infective treatment, including but not limited to tuberculosis, HBV or HCV infection, HIV infection, or CMV infection.
* Major surgical procedures within the preceding three months.
* Hypersensitivity or intolerance to Firsekibart; individuals with known hypersensitivity to Chinese hamster ovary (CHO) cell-derived products should also be excluded (Firsekibart is a recombinant monoclonal antibody with potential residual CHO expression risk).
* Pregnancy, planned pregnancy, or lactation.
* Use of biological agents within 3 months prior to enrolment, including but not limited to CD20 monoclonal antibodies (e.g., rituximab), B-lymphocyte stimulatory factor inhibitors (e.g., belimumab, telitacicept), or TNF-α inhibitors (e.g., adalimumab, infliximab).
* Receipt within 3 months prior to enrolment of high-dose glucocorticoids (prednisolone or equivalent ≥60mg qd), plasma exchange, IVIG, or oral/intravenous cyclophosphamide.
* Individuals who have received live attenuated vaccines (e.g., varicella, herpes zoster, intranasal influenza vaccines) within 3 months prior to enrolment, or who plan to receive live vaccines during the study period.
* Any condition deemed by the investigator to potentially prevent the subject from completing the study or pose a significant risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients achieving an BICLA response at the end of 12 weeks | From enrollment to the end of treatment at 12 weeks
  The BICLA response was defined as a reduction of all severe (BILAG-2004 A) or moderately severe (BILAG-2004 B) disease activity at baseline to lower levels (BILAG-2004 B, C, or D and C or D, respectively) and no worsening in other organ systems (with worsening defined as ≥1 new BILAG-2004 A item or ≥2 new BILAG-2004 B items); no worsening in disease activity, as determined by the SLEDAI-2K score (no increase from baseline) and by the PGA score (no increase of ≥0.3 points from baseline)

SECONDARY OUTCOMES:
the percentage of patients achieving an BICLA response at the end of 24 weeks | From enrollment to the end of treatment at 24 weeks
  The BICLA response was defined as a reduction of all severe (BILAG-2004 A) or moderately severe (BILAG-2004 B) disease activity at baseline to lower levels (BILAG-2004 B, C, or D and C or D, respectively) and no worsening in other organ systems (with worsening defined as ≥1 new BILAG-2004 A item or ≥2 new BILAG-2004 B items); no worsening in disease activity, as determined by the SLEDAI-2K score (no increase from baseline) and by the PGA score (no increase of ≥0.3 points from baseline)
the percentage of patients achieving SRI-4 response at the end of 12 weeks. | From enrollment to the end of treatment at 12 weeks
  The SRI-4（SLE Responder Index-4） response was defined as a reduction of at least 4 points in SLEDAI score compared with the baseline level, no new British Isles Lupus Assessment Group (BILAG) A organ domain score or no more than one new BILAG B organ domain score, and no worsening in the Physician's Global Assessment (PGA) (<0.3 points worsening from the baseline level).
the percentage of patients achieving SRI-4 response at the end of 24 weeks. | From enrollment to the end of treatment at 24 weeks
  The SRI-4（SLE Responder Index-4） response was defined as a reduction of at least 4 points in SLEDAI score compared with the baseline level, no new British Isles Lupus Assessment Group (BILAG) A organ domain score or no more than one new BILAG B organ domain score, and no worsening in the Physician's Global Assessment (PGA) (<0.3 points worsening from the baseline level).
Changes from baseline in SLEDAI at 24 weeks | From enrollment to the end of treatment at 24 weeks
  SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index, with a score of 0-6 representing mild disease activity, 7-12 representing moderate disease activity, and 12-16 representing severe disease activity
Changes from baseline in SLEDAI at 12 weeks | From enrollment to the end of treatment at 12 weeks
  SLEDAI stands for Systemic Lupus Erythematosus Disease Activity Index, with a score of 0-6 representing mild disease activity, 7-12 representing moderate disease activity, and 12-16 representing severe disease activity
Changes from baseline in PGA at 24 weeks | From enrollment to the end of treatment at 24 weeks
  PGA stands for Physician's Global Assessment (PGA ) . It is used to assess the activity of systemic lupus erythematosus on a scale ranging from 0 to 3, where 0 indicates no disease activity and 3 indicates the most severe disease activity.
Changes from baseline in PGA at 12 weeks | From enrollment to the end of treatment at 12 weeks
  PGA stands for Physician's Global Assessment (PGA ) . It is used to assess the activity of systemic lupus erythematosus on a scale ranging from 0 to 3, where 0 indicates no disease activity and 3 indicates the most severe disease activity.
Changes from baseline of the SJC and TJC at 24 weeks | From enrollment to the end of treatment at 24 weeks
  Swollen Joint Count(SJC) and Tender Joint Count(TJC) indicate the number of swollen and tender joints in 28 joints, respectively. 28 joints refer to both shoulders, both elbows, both wrists, both knees, 10 metacarpophalangeal joints, and 10 proximal interphalangeal joints, which ranging from 0 to 28, the higher value means more serious disease activity.
Changes from baseline of the SJC and TJC at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Swollen Joint Count(SJC) and Tender Joint Count(TJC) indicate the number of swollen and tender joints in 28 joints, respectively. 28 joints refer to both shoulders, both elbows, both wrists, both knees, 10 metacarpophalangeal joints, and 10 proximal interphalangeal joints, which ranging from 0 to 28, the higher value means more serious disease activity.
Changes from baseline of the levels of Erythrocyte Sedimentation Rate (ESR) at 24 weeks | From enrollment to the end of treatment at 24 weeks
  The erythrocyte sedimentation rate (ESR) is used to indicate the level of inflammation. In this study, the normal range is 0-15 mm/h. A value exceeding the upper limit of normal indicates an elevated level of inflammation, with higher values suggesting a greater degree of inflammation.
Changes from baseline of the levels of Erythrocyte Sedimentation Rate (ESR) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  The erythrocyte sedimentation rate (ESR) is used to indicate the level of inflammation. In this study, the normal range is 0-15 mm/h. A value exceeding the upper limit of normal indicates an elevated level of inflammation, with higher values suggesting a greater degree of inflammation.
Changes from baseline of the CLASI score at 24 weeks | From enrollment to the end of treatment at 24 weeks
  The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) was used in this study to evaluate disease activity and lesion severity in cutaneous SLE involvement. Scores of 0-9 indicate mild disease, 10-20 moderate disease, and 21-70 severe disease.
Changes from baseline of the CLASI score at 12 weeks | From enrollment to the end of treatment at 12 weeks
  The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) was used in this study to evaluate disease activity and lesion severity in cutaneous SLE involvement. Scores of 0-9 indicate mild disease, 10-20 moderate disease, and 21-70 severe disease.
Changes from baseline of the levels of C-Reaction Protein (CRP) at 24 weeks | From enrollment to the end of treatment at 24 weeks
  The c-reaction protein (CRP) is used to indicate the level of inflammation. In this study, the normal range is 0-10 mg/L. A value exceeding the upper limit of normal indicates an elevated level of inflammation, with higher values suggesting a greater degree of inflammation.
Changes from baseline of the levels of C-Reaction Protein (CRP) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  The c-reaction protein (CRP) is used to indicate the level of inflammation. In this study, the normal range is 0-10 mg/L. A value exceeding the upper limit of normal indicates an elevated level of inflammation, with higher values suggesting a greater degree of inflammation.